CLINICAL TRIAL: NCT00139737
Title: Open Extension Study Evaluating the Safety and Tolerability of Oral Ziprasidone in the Treatment of Subjects Who Have Successfully Completed a Previous Ziprasidone Study
Brief Title: Extension Study: Evaluating the Safety of Oral Ziprasidone in the Treatment of Subjects With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281061
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Results first posted 2010-07-14 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia
Keywords: Open-label extension Ziprasidone study in Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ziprasidone — 20mg capsules BID, 40mg capsules BID, 60mg BID or 80mg BID until drug commercialisation in Italy.
  Other Names: Geodon, Zeldox

SUMMARY:
To provide treatment to eligible subjects who have successfully completed one of the following phase III ziprasidone studies, A1281028, A1281044, A1281045 (NCT00136994) or A1281088 (NCT00143351).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have successfully completed a ziprasidone clinical study
* Patients not hospitalised in an acute psychiatric service
* Written, informed consent to participation.
* Female patients of at risk of pregnancy must avoid to remain pregnant; an adequate method of contraception (intrauterine device, implanted contraceptive, oral contraceptive or condom) must be initiated or continued

Exclusion Criteria:

Psychiatric:

* Subjects at immediate risk of committing harm to self or others
* Subjects requiring concurrent treatment with non-study antipsychotic agents
* Subjects requiring treatment with antidepressants or mood stabilizers
* General:
* Subjects with a history of clinically significant and/or currently relevant hematological, renal (including single kidney), hepatic, gastrointestinal, endocrine (except for current adequately treated hypo- or hyperthyroidism), pulmonary (excluding chronic bronchitis, mild emphysema or chronic obstructive pulmonary disease), dermatological, oncological, or neurological disease, excluding tardive dyskinesia but including all forms of epilepsy (febrile convulsions in childhood acceptable). The only subjects with known prior malignant disease who are eligible are those with cured prior skin cancer (excluding melanoma). Controlled Type II diabetes (glucose < 180 mg/100 ml at screening and baseline with dietary or oral hypoglycemic treatment) will not be considered a significant medical illness and would not exclude a subject from the study
* Acute or chronic heart disease
* Clinically significant ECG abnormalities
* Subjects with QTc >= 500 msec (subjects with QTc >= 450 msec and < 500 msec should be discussed with the cardiologist who is responsible for all of the centers involved)
* Concomitant treatment with medications that prolong QTc interval (please review prescribing information of other treatments)
* Subjects with serum K+ or Mg++ outside the normal range
* Subject with any confirmed laboratory values that deviate from the upper or lower limits of normal prior to study entry, except for clinically insignificant deviations as determined by investigator
* Known serological evidence of HIV, or acute or chronic hepatitis (with transaminase levels higher than three times upper limit)
* Pregnant or lactating women
* Subjects who intend to donate blood or blood products during the 4 weeks prior to the study, during the study or in the 30 days after the study ends
* Subjects unable or unlikely to follow the study protocol
* Subjects with a history of neuroleptic malignant syndrome developing from the administration of antipsychotic compounds
* Known hypersensitivity to ziprasidone or lactose

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 344 (Actual)
Dates: Start 2002-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (76):
- Italy (76):
  - Pfizer Investigational Site, Sora, Frosinone
  - Pfizer Investigational Site, Parma, PR
  - Pfizer Investigational Site, Acri, CS
  - Pfizer Investigational Site, Arezzo
  - Pfizer Investigational Site, Arona (No)
  - Pfizer Investigational Site, Bassano del Grappa
  - Pfizer Investigational Site, Bisceglie (BA)
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Bolzano
  - Pfizer Investigational Site, Brindisi
  - Pfizer Investigational Site, Cagliari
  - Pfizer Investigational Site, Casalecchio Di Reno BO
  - Pfizer Investigational Site, Caserta
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Cefalu' (Pa)
  - Pfizer Investigational Site, Cesena FO
  - Pfizer Investigational Site, Chiari (Bs)
  - Pfizer Investigational Site, Cremona
  - Pfizer Investigational Site, Crotone
  - Pfizer Investigational Site, Cuneo
  - Pfizer Investigational Site, Dolo (Ve)
  - Pfizer Investigational Site, Empoli
  - Pfizer Investigational Site, Enna
  - Pfizer Investigational Site, Fano (PS)
  - Pfizer Investigational Site, Formia (LT)
  - Pfizer Investigational Site, Frattaminore (NA)
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Genzano (RM)
  - Pfizer Investigational Site, Giarre, CT
  - Pfizer Investigational Site, Guardiagrele (CH)
  - Pfizer Investigational Site, Lamezia Terme
  - Pfizer Investigational Site, Lecce
  - Pfizer Investigational Site, Livorno
  - Pfizer Investigational Site, L’Aquila
  - Pfizer Investigational Site, Matera
  - Pfizer Investigational Site, Melzo (MI)
  - Pfizer Investigational Site, Merano (BZ)
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Montebelluna (TV)
  - Pfizer Investigational Site, Montecchio Maggiore (VI)
  - Pfizer Investigational Site, Montevarchi (AR)
  - Pfizer Investigational Site, Monza MI
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Nocera Inferiore, SA
  - Pfizer Investigational Site, Noto
  - Pfizer Investigational Site, Novi Ligure, AL
  - Pfizer Investigational Site, Orbassano, to
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Partinico (Pa)
  - Pfizer Investigational Site, Passirana Di Rho (Mi)
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Pordenone
  - Pfizer Investigational Site, Portogruaro (Ve)
  - Pfizer Investigational Site, Puglianello (BN)
  - Pfizer Investigational Site, Ragusa
  - Pfizer Investigational Site, Reggio Calabria
  - Pfizer Investigational Site, Rivoli, to
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Salerno
  - Pfizer Investigational Site, San Benedetto Del Tronto, AP
  - Pfizer Investigational Site, San Giorgio Di Piano BO
  - Pfizer Investigational Site, San Marco in Lamis FG
  - Pfizer Investigational Site, Sant'Arsenio (SA)
  - Pfizer Investigational Site, Sassari
  - Pfizer Investigational Site, Senigallia, AN
  - Pfizer Investigational Site, Spoleto (PG)
  - Pfizer Investigational Site, Taranto
  - Pfizer Investigational Site, Tivoli (RM)
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Treviso
  - Pfizer Investigational Site, Udine
  - Pfizer Investigational Site, Verona
  - Pfizer Investigational Site, Viareggio

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281061&StudyName=Extension%20Study%3A%20Evaluating%20the%20Safety%20of%20Oral%20Ziprasidone%20in%20the%20Treatment%20of%20Subjects%20with%20Schizophrenia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study enrolled eligible subjects with schizophrenia who had successfully completed a previous Phase 3 ziprasidone study (A1281028, A1281044 or A1281045 [NCT00136994]), allowing enrolled subjects to continue treatment with ziprasidone for at least 1 year or until the drug became commercially available.
Groups:
- Ziprasidone: Ziprasidone treatment was continued at the same dose used in the previous protocol with subsequent dose adjustments within 20-40-60-80 mg twice daily according to investigator's opinion on clinical status of subject. The maximum total daily oral dose allowed was 160 mg.
Period: Overall Study
Arm/Group | Ziprasidone
Started | 344
Received Treatment | 331
Completed | 3
Not Completed | 341
Not completed — Withdrawal by Subject | 190
Not completed — Adverse Event | 58
Not completed — Lack of Efficacy | 40
Not completed — Lost to Follow-up | 8
Not completed — Death | 3
Not completed — Laboratory Abnormality | 2
Not completed — Protocol Violation | 18
Not completed — Withdrew During Screening Phase | 8
Not completed — Did Not Meet Entrance Criteria | 1
Not completed — Screened, Not Treated | 13

BASELINE CHARACTERISTICS:
Arm/Group | Ziprasidone
Number analyzed (Participants) | 331
Age, Customized [Number; unit: Participants]
  18-44 years | 238
  45-64 years | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 193

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: All observed or volunteered treatment-emergent AEs and SAEs regardless of treatment group or suspected causal relationship to the investigational product were reported.
Time Frame: Baseline up to 72 months
Population: Safety Analysis Set = All subjects who took at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 331
Participants
  AEs | 177
  SAEs | 32

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 32/331
Other Adverse Events (participants affected / at risk) | 177/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=331)
Myocardial ischaemia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Irritability (General disorders) | 2
Accident (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epilepsy (Nervous system disorders) | 1
Mental impairment (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 2
Alcohol abuse (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Dysphoria (Psychiatric disorders) | 1
Hypomania (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 14
Suicide attempt (Psychiatric disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=331)
Arrhythmia (Cardiac disorders) | 1
Bundle branch block right (Cardiac disorders) | 2
Conduction disorder (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Goitre (Endocrine disorders) | 1
Hyperprolactinaemia (Endocrine disorders) | 5
Hyperthyroidism (Endocrine disorders) | 1
Diplopia (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 6
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
Influenza like illness (General disorders) | 1
Irritability (General disorders) | 1
Pyrexia (General disorders) | 3
Swelling (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Cystitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gingival abscess (Infections and infestations) | 1
Helicobacter gastritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 7
Labyrinthitis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Drug administration error (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood prolactin increased (Investigations) | 5
Electrocardiogram QT prolonged (Investigations) | 46
Electrocardiogram abnormal (Investigations) | 11
Glycosylated haemoglobin increased (Investigations) | 1
Laboratory test abnormal (Investigations) | 1
Lipids increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Weight decreased (Investigations) | 5
Weight increased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Akathisia (Nervous system disorders) | 2
Autism (Nervous system disorders) | 1
Cogwheel rigidity (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Extrapyramidal disorder (Nervous system disorders) | 6
Headache (Nervous system disorders) | 11
Hemiparesis (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Psychomotor hyperactivity (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 11
Tremor (Nervous system disorders) | 3
Affect lability (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 11
Anxiety (Psychiatric disorders) | 15
Apathy (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 11
Disinhibition (Psychiatric disorders) | 2
Dysphoria (Psychiatric disorders) | 1
Elevated mood (Psychiatric disorders) | 1
Euphoric mood (Psychiatric disorders) | 2
Hallucination (Psychiatric disorders) | 2
Hallucination, auditory (Psychiatric disorders) | 2
Hypochondriasis (Psychiatric disorders) | 1
Hypomania (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 21
Libido decreased (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Paranoia (Psychiatric disorders) | 1
Psychiatric symptom (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 6
Restlessness (Psychiatric disorders) | 2
Schizophrenia (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 5
Tension (Psychiatric disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Ejaculation disorder (Reproductive system and breast disorders) | 1
Ejaculation failure (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2
Gynaecomastia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.